CLINICAL TRIAL: NCT02921971
Title: Efficacy and Safety of SAR156597 in the Treatment of Diffuse Cutaneous Systemic Sclerosis (dcSSc): A Randomized, Double-blind, Placebo-controlled, 24-week, Proof of Concept Study
Brief Title: Effectiveness and Safety of SAR156597 in Treating Diffuse Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT14604; 2016-001028-80 (EudraCT Number); U1111-1179-4690 (Other: UTN)
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Results first posted 2022-02-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo (for SAR156597), single subcutaneous (SC) injection once in a week (QW) up to Week 24.
  Interventions: Drug: Placebo
- SAR156597 (Experimental): SAR156597 200 milligram (mg), single SC injection QW up to Week 24.
  Interventions: Drug: SAR156597

INTERVENTIONS:
Drug: SAR156597 — Pharmaceutical form: Solution Route of administration: Subcutaneous
  Other Names: Romilkimab
  Arms: SAR156597
Drug: Placebo — Pharmaceutical form: Solution Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate, in comparison with placebo, the efficacy of SAR156597 administered subcutaneously for 24 weeks on skin fibrosis in participants with diffuse cutaneous systemic sclerosis (dcSSc).

Secondary Objectives:

* To evaluate the efficacy of SAR156597 compared to placebo on physical/functional disability in participants with dcSSc.
* To evaluate the efficacy of SAR156597 compared to placebo on respiratory function of participants with dcSSc.
* To evaluate the safety profile of SAR156597 compared to placebo in participants with dcSSc.
* To evaluate the potential for immunogenicity (anti-drug antibodies response) of SAR156597 in participants with dcSSc.
* To evaluate the pharmacokinetics (trough plasma concentrations) of SAR156597 administered subcutaneously for 24 weeks.

DETAILED DESCRIPTION:
The total study duration per participant was 39 weeks; consisting of a 4-week screening, a 24-week of study treatment period, and an 11-week follow-up with no study drug treatment.

ELIGIBILITY:
Inclusion criteria :

* Systemic Sclerosis (SSc) according to the American College of Rheumatology/The European League against Rheumatism (ACR/EULAR) 2013 criteria.
* Diffused cutaneous form of SSc according to Leroy's criteria.
* Able and willing to sign the written informed consent form with comprehension of its contents and complied with the requirements of the study protocol.

Exclusion criteria:

* Aged less than (<) 18 years of age.
* Disease duration for greater than (>) 36 months from time of first non-Raynaud's phenomenon manifestation.
* Modified Rodnan Skin Score <10 or >35 at screening and baseline visits.
* History of vasculitis, active or in remission.
* Diagnosis of connective tissue diseases (other than SSc) or overlap syndrome (eg, polymyositis/scleroderma).
* Positive Human Immunodeficiency Virus (HIV) serology or a known history of HIV infection, active or in remission.
* Abnormal hepatitis B and/or hepatitis C tests indicative of active or chronic infection:
* Abnormal Hepatitis B tests: Positive hepatitis B surface antigen (HBsAg) OR positive total hepatitis B core antibody (HBcAb) with negative hepatitis B surface antibody (HBsAb) OR positive total HBcAb with positive HBsAb and presence of hepatitis B virus deoxyribonucleic acid.
* Abnormal Hepatitis C tests: Positive anti-hepatitis C virus antibody (HCV Ab) and positive HCV ribonucleic acid.
* Positive or 2 confirmed indeterminate Quantiferon-tuberculosis Gold tests at screening (regardless of prior treatment status).
* Serious infection (eg, pneumonia, pyelonephritis) within 4 weeks of screening, infection requiring hospitalization or intravenous antibiotics within 4 weeks of screening or chronic bacterial infection (eg, osteomyelitis).
* History of anaphylaxis to any biologic therapy.
* Evidence of any clinically significant, severe or unstable, acute or chronically progressive, uncontrolled infection or medical condition (eg, cerebral, cardiac, pulmonary, renal, hepatic, gastrointestinal or neurologic other than SSc or SSc-interstitial lung disease) or previous, active or pending surgical disorder, or any condition that may affect participant safety in the judgment of the Investigator.
* At screening, the percent (%) predicted forced vital capacity was less than or equal to (<=75) % and % predicted carbon monoxide diffusing lung capacity after hemoglobin correction is <=40%.
* History of heart failure (including acutely decompensated in the setting of preserved ejection fraction), left ventricular ejection fraction <= 45%, coronary artery disease, angina, myocardial infarction, ischemic cardiomyopathy and/or hypertrophic cardiomyopathy.
* Any prior history of malignancy or active malignancy, including lymphoproliferative diseases (except successfully-treated carcinoma in-situ of the cervix, non-metastatic squamous cell carcinoma or basal cell carcinoma of the skin) within 5 years prior to baseline.
* Ischemic electrocardiogram (ECG) changes (except those not supported by the findings of a left heart catheterization performed in the last year) and/or other clinically significant ECG findings. (All abnormal ECG finding were reviewed and confirmed by a local cardiologist).
* High dose steroids (>10 mg/day prednisolone equivalent); or change in steroid dose within 4 weeks prior to randomization (or baseline visit); or expected changes during the course of the study.
* Previous treatment with rituximab within 12 months prior to screening.
* Previous treatment with bone marrow transplantation, total lymphoid irradiation or ablative ultra-high dose cyclophosphamide.
* Treatment with high dose immunosuppressive drug (eg, cyclophosphamide >1 mg/kilogram (kg) oral/day or >750 mg intravenous (IV)/month; azathioprine >100 mg/day; methotrexate >15 mg/week; mycophenolate mofetil >2 gram (g)/day) within 3 months of screening or change in dose within 4 weeks prior to randomization (or baseline visit); or expected changes in dose during the course of the study.
* Treatment with etanercept, cyclosporine A, IV immunoglobulin, rapamycin, D-penicillamine, tyrosine kinase inhibitors within 4 weeks of screening or antithymocyte globulin within 6 months of screening.
* Treatment with infliximab, certolizumab, golimumab, abatacept, or adalimumab, tocilizumab within 8 weeks of screening or anakinra within 1 week of screening.
* Treatment with any investigational drug within 1 month of screening, or 5 half-lives, if known (whichever was longer).
* Abnormal laboratory tests at screening:
* Alanine transaminase or aspartate transaminase >2 times upper limit of normal range;
* Hemoglobin <11 g/100 milliliter (mL) for male and <10 g/100 mL for female;
* Neutrophils <1500/mm^3 (except <1000/mm^3 for those of African descent);
* Platelets <100 000/mm^3;
* Creatinine greater than or equal to (>=)150 micromole/Liter (mcgmol/L).
* Current history of substance and/or alcohol abuse.
* Any condition or circumstance that would preclude the participant from following and completing protocol requirements, in the opinion of the Investigator.
* Pregnant or breastfeeding woman.
* Women who were of childbearing potential not protected by highly-effective contraceptive method(s) of birth control, and/or who were unwilling or unable to be tested for pregnancy.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (44):
- United States (4):
  - Investigational Site Number 8400006, San Francisco, California
  - Investigational Site Number 8400005, Washington D.C., District of Columbia
  - Investigational Site Number 8400002, Cleveland, Ohio
  - Investigational Site Number 8400007, Houston, Texas
- Argentina (4):
  - Investigational Site Number 0320003, Buenos Aires
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320005, Capital Federal
  - Investigational Site Number 0320001, San Miguel de Tucumán
- Belgium (2):
  - Investigational Site Number 0560001, Ghent
  - Investigational Site Number 0560002, Leuven
- Investigational Site Number 2330001, Tallinn, Estonia
- France (3):
  - Investigational Site Number 2500003, Montpellier
  - Investigational Site Number 2500004, Paris
  - Investigational Site Number 2500002, Strasbourg
- Germany (4):
  - Investigational Site Number 2760003, Bad Nauheim
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760002, Cologne
  - Investigational Site Number 2760004, Ulm
- Italy (4):
  - Investigational Site Number 3800004, Genova
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800005, Milan
  - Investigational Site Number 3800006, Orbassano
- Mexico (4):
  - Investigational Site Number 4840001, Chihuahua City
  - Investigational Site Number 4840005, Guadalajara
  - Investigational Site Number 4840002, Guadalajara
  - Investigational Site Number 4840003, Monterrey
- Poland (3):
  - Investigational Site Number 6160001, Poznan
  - Investigational Site Number 6160002, Warsaw
  - Investigational Site Number 6160003, Wroclaw
- Romania (5):
  - Investigational Site Number 6420003, Bucharest
  - Investigational Site Number 6420004, Bucharest
  - Investigational Site Number 6420005, Bucharest
  - Investigational Site Number 6420001, Cluj-Napoca
  - Investigational Site Number 6420002, Târgu Mureş
- Russia (5):
  - Investigational Site Number 6430002, Kemerovo
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430003, Ufa
- Ukraine (4):
  - Investigational Site Number 8040001, Kyiv
  - Investigational Site Number 8040002, Kyiv
  - Investigational Site Number 8040004, Kyiv
  - Investigational Site Number 8040003, Kyiv
- Investigational Site Number 8260001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Allanore Y, Wung P, Soubrane C, Esperet C, Marrache F, Bejuit R, Lahmar A, Khanna D, Denton CP; Investigators. A randomised, double-blind, placebo-controlled, 24-week, phase II, proof-of-concept study of romilkimab (SAR156597) in early diffuse cutaneous systemic sclerosis. Ann Rheum Dis. 2020 Dec;79(12):1600-1607. doi: 10.1136/annrheumdis-2020-218447. Epub 2020 Sep 22. PMID 32963047

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 13 countries. A total of 97 participants were involved in the study from 21 December 2016 to 01 April 2019.
Pre-assignment Details: Participants were randomized in 1:1 ratio (placebo and SAR156597). Randomization was stratified based upon the participant's medical history of systemic sclerosis (SSc) associated interstitial lung disease (SSc-ILD) (yes or no). Assignment was done by Interactive Voice Response System (IVRS).
Period: Overall Study
Arm/Group | Placebo | SAR156597
Started | 49 | 48
Completed | 43 | 44
Not Completed | 6 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 3 | 1
Not completed — Other than specified above | 2 | 1

BASELINE CHARACTERISTICS:
Population: The analysis was performed on all randomized population.
Groups:
- Placebo: Placebo (for SAR156597), single SC injection QW up to Week 24.
- SAR156597: SAR156597 200 mg, single SC injection QW up to Week 24.
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR156597 | Total
Number analyzed (Participants) | 49 | 48 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.1) | 52.3 (10.8) | 49.7 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 2 | 4
  White | 45 | 45 | 90
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: units on a scale] — mRSS: an accepted clinical measure of the skin thickness (fibrosis). Investigator physicians or qualified medical personnel assessed the thickening of skin in 17 skin sites, including fingers, hands, forearms, arms, feet, legs and thighs, face, chest and abdomen. Each skin site was rated on a 0-3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness. Total mRSS (sum of individual scores) ranged from 0 (normal skin) to 51 (severe thickening in all 17 areas), where higher score indicated more severity of skin thickening/worst outcome.
  units on a scale | 20.6 (7.0) | 20.5 (6.1) | 20.6 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Rodnan Skin Score to Week 24
Description: mRSS, an accepted clinical measure of the skin thickness (fibrosis). Investigator physicians or qualified medical personnel assessed the thickening of skin in 17 skin sites including fingers, hands, forearms, arms, feet, legs and thighs, face, chest and abdomen. Each skin site was rated on a 0-3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness and 3 = severe thickness. Total mRSS ranged from 0 (no thickening) to 51 (severe thickening in all 17 areas), where higher score indicated more severity of skin thickening/worst outcome.
Time Frame: Baseline, Week 24
Population: Analysis was performed on the intent to treat (ITT) population which included all randomized participants and were analyzed according to the treatment group allocated by randomization. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR156597
Number analyzed (Participants) | 48 | 47
score on a scale | -2.45 (0.85) | -4.76 (0.86)
Statistical Analysis 1: Comparison: Placebo vs SAR156597; Analysis was performed using mixed model repeated measures (MMRM) model. The model included fixed categorical effects of treatment group, randomization strata as per IVRS, timepoint, treatment-by-timepoint and strata-by-timepoint interactions, as well as the continuous fixed covariate of baseline and baseline-by-timepoint interactions; Test type: Superiority; p = 0.0291, Mixed-effect model with repeated measure — Above p-value is one-sided p-value. Threshold for significance is at 0.05 level; Least square (LS) Mean difference = -2.31, 95% CI 2-sided [-4.71 to 0.08], Standard Error of Mean 1.21

2. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) Score to Week 24
Description: HAQ-DI assessed the degree of difficulty participants experienced in 8 daily living activity domains during past week: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Each activity category consisted of 2-3 items. For each items, level of difficulty was scored from 0-3 (0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do). Overall HAQ-DI score was computed as the sum of domain scores divided by the number of domains answered, providing a score from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability.
Time Frame: Baseline, Week 24
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | SAR156597
Number analyzed (Participants) | 48 | 47
score on a scale | -0.12 (0.08) | -0.09 (0.08)

3. Secondary Outcome: Change From Baseline in Mean Observed Forced Vital Capacity (FVC) Level to Week 24
Description: FVC was the total amount of air (in liters) exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying ILD. Change from Baseline was calculated by subtracting Baseline value from Week 24 value.
Time Frame: Baseline, Week 24
Population: Analysis was performed on the ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | SAR156597
Number analyzed (Participants) | 47 | 47
liters | -0.08 (0.04) | -0.01 (0.04)

4. Secondary Outcome: Change From Baseline in Mean Observed Diffusing Lung Capacity for Carbon Monoxide (DLco) to Week 24
Description: DLco is a measurement of the ability of the lungs to transfer gases from the air to the blood. Participant breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participant hold the breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine amount of the tracer gas absorbed during the breath.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimoles per minute per kilopascal
Arm/Group | Placebo | SAR156597
Number analyzed (Participants) | 46 | 47
millimoles per minute per kilopascal | -0.27 (0.10) | -0.12 (0.10)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from the signature of the informed consent form until the end of the study, regardless of seriousness or relationship to investigational medicinal product (IMP). Reported treatment-emergent adverse events (TEAEs) and deaths were AEs that developed or worsened or became serious during the TEAE period, defined as the time from the first administration of the IMP up to 12 weeks (84 days) from the last dose of IMP (i.e. up to 36 weeks).
Description: Analysis was performed on safety population which included all participants who received at least 1 dose or part of a dose of the study drug and were analyzed according to the treatment actually received.
Groups:
- SAR156597: SAR156597 200 mg single SC injection QW up to Week 24.
Arm/Group | Placebo | SAR156597
All-Cause Mortality (participants affected / at risk) | 1/49 | 1/48
Serious Adverse Events (participants affected / at risk) | 5/49 | 4/48
Other Adverse Events (participants affected / at risk) | 27/49 | 31/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | SAR156597 (N=48)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Intestinal Pseudo-Obstruction (Gastrointestinal disorders) | 1 (3) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Acute (Infections and infestations) | 1 (1) | 0 (0)
Echocardiogram Abnormal (Investigations) | 1 (1) | 0 (0)
Scleroderma Renal Crisis (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=49) | SAR156597 (N=48)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 7 (8)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 3 (3)
Cystitis (Infections and infestations) | 2 (2) | 3 (3)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6)
Oral Herpes (Infections and infestations) | 1 (1) | 5 (7)
Pharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 1 (1) | 4 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (4)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 15 (23) | 8 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2017-08-09): https://cdn.clinicaltrials.gov/large-docs/71/NCT02921971/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT02921971/SAP_001.pdf